CLINICAL TRIAL: NCT01123200
Title: An In-home Study of Brain Computer Interfaces
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jane Huggins, PhD, Research Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: J0002
Record Dates: First submitted 2010-05-04; First posted 2010-05-14 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Brain-Computer Interfaces

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brain Computer Interface In-Home Use (Other)
  Interventions: Device: Brain Computer Interface for Wheelchair Tilt Control

INTERVENTIONS:
Device: Brain Computer Interface for Wheelchair Tilt Control — Patients will be given the BCI for use in-home, as long as they use the BCI at least 10 hours per week and complete monthly performance assessment sessions.

SUMMARY:
The investigators are developing a tool to help people who are severely paralyzed. This tool is called a brain-computer interface (BCI). BCIs can connect to computers or other electronic devices.

This study allows a person with ALS to communicate, control their wheelchair tilt and perform other tasks using a BCI, thus increasing their independence.

DETAILED DESCRIPTION:
This small-scale study of the feasibility of a BCI to operate the tilt position of a power wheelchair was also designed to determine the conditions and support structures necessary for use of a BCI in the home. In this study, people with Amyotrophic Lateral Sclerosis (ALS) will have a BCI in their home. They will receive training in order to operate and maintain the BCI. The BCI will allow them to access at least one task of primary interest to them. Task may include communication, computer access, control of assistive technology, or control of wheelchair seat position. Data concerning the use of the BCI will be collected throughout the study. Custom installations will be made for each participant to connect to their wheelchair and provide communication options if needed. Each installation is expected to be a unique prototype because of the differing control requirements for the individual wheelchairs in use by the participants.

We intended to enroll six participants, but were only able to enroll one.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Presently having difficulty communicating or operating the controls for assistive technology or likely to have difficulty in the next six months.
* Able to see the BCI display
* Able to understand and remember instructions concerning participation.
* Live in an environment that can accommodate the wheelchair portable BCI host computer
* Expected to live in the same physical environment for at least 6 months.
* Has family and caregiver(s) who are supportive of participation in this research.
* Has a primary caregiver who is technically capable, willing to learn the setup and operation of the BCI system, and likely to remain with the subject for at least 6 months.
* Has been shown to be able to use a BCI (in an experimental session under another IRB, e.g. HUM 00012968).
* Has a clear understanding of the shortcomings of the present state of BCI technology

Exclusion Criteria:

* Open head lesions or a history of problems with skin breakdown on the head that may be aggravated by repeated application of electrodes.
* Inability to communicate well enough to give informed consent.
* History of photo-sensitive epilepsy
* Known significant cognitive deficits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Huggins, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brain Computer Interface In-Home Use
Started | 1
Completed | 0
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Brain Computer Interface In-Home Use
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Duration of BCI Usage by Persons With ALS.
Description: Number of months of BCI usage by each participant.
Time Frame: Monthly measurements for a period of up to 18 months.
Measure: Mean (Full Range); unit: months
Arm/Group | Brain Computer Interface In-Home Use
Number analyzed (Participants) | 1
months | 5 [5 to 5]

2. Secondary Outcome: Changes in Accuracy of BCI for Controlling Devices and Text
Description: Changes in Accuracy Percentage (i.e., cumulative correct selections per month divided by the cumulative number of intended sections per month). Looking for trends over each 6 month period.
Time Frame: 6 months, 12 months, 18 months
Population: The first six month period was not completed by any participant so accuracy data for six months could not be analyzed.
Arm/Group | Brain Computer Interface In-Home Use
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Brain Computer Interface In-Home Use
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brain Computer Interface In-Home Use (N=1)
Unexpected wheelchair movement (Product Issues) | 1 (1) — After the BCI was shut down and disconnected, the wheelchair reportedly moved without the user operating the controls. The movement was brief and no injury occurred.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No